CLINICAL TRIAL: NCT03147183
Title: Kinetic Study of CD8+ CMV-specific Cellular Immunity in Renal Transplant Patients After Receiving Thymoglobulin
Status: Completed | Type: Observational
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Responsible Party: Sponsor
Other Study IDs: FIB-TIM-2015-01
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Renal Transplant Infection
MeSH Terms: interventions — thymoglobulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- candidates for renal transplant
  Interventions: Drug: Thymoglobulin

INTERVENTIONS:
Drug: Thymoglobulin — This study will use non-probability, convenience sampling from patients kidney transplants who receive induction immunosuppressive therapy with thymoglobulin

SUMMARY:
Renal transplant candidates who have CMV-specific, CD8+ T-cells, are CMV-seropositive and carry HLA-A1 and/ or HLA- A2 alleles have a high probability to maintain this type of immunity during the three first months after the transplant, despite induction immunosuppressive therapy (thymoglobulin).

ELIGIBILITY:
Inclusion Criteria:

1. Renal transplant recipients with CMV-positive serology.
2. Patients with pre-transplant, CMV-specific CD8+ T cell-mediated immunity, i.e. IFNγ levels ≥0.2 UI/mL (QF-CMV Reactive).
3. Adults over 18 years of age.
4. Patients receiving induction therapy with thymoglobulin (at least a cumulative dosage of 1mg/kg).
5. Patients receiving prophylaxis with valganciclovir (900 mg/day, adjusted to kidney function) until day 90 after transplant.
6. Patients who signed an informed consent

Exclusion Criteria:

1. Multivisceral transplantation, including pancreas-kidney transplantation.
2. HIV infected patients.
3. Patients who cannot comply with the monitoring protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are candidates for renal transplant and who fulfil the clinical criteria established by the participating institutions to receive induction immunosuppressive therapy. Participating institutions may include centers from the Spanish Network for Research in Infectious Diseases (REIPI, Transplantation Program) as well as other centers outside the network.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2016-08-09 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
CMV-specific, CD8+ T-cell immunity | 18 months
  Percentage of patients with CMV-specific, CD8+ T-cell immunity at any of the established time points for monitorization. "CMV-specific, CD8+ T-cell immunity" will be defined as production of IFNγ ≥0.2 UI/mL (QF-CMV Reactive).

CONTACTS AND LOCATIONS:
Locations (1):
- Hosìtal Universitario Reina Sofia, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No